CLINICAL TRIAL: NCT04210596
Title: A Multicenter Randomized Controlled Study Comparing Connective Tissue Graft with Collagen Matrix to Re-establish Convexity At the Buccal Aspect of Single Dental Implants
Brief Title: Connective Tissue Graft Versus Collagen Matrix
Acronym: BC-5303
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-178; BOF.STG.2019.0004.01 (Other Grant/Funding Number: BOF Ghent University); 18-178 (Other Grant/Funding Number: Osteology Foundation)
Record Dates: First submitted 2019-10-07; First posted 2019-12-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Buccal Soft Tissue Profile (BSP)
Keywords: connective tissue graft; collagen matrix; dental implant, single tooth; volumetric analysis

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled study with 2 treatment arms (control: connective tissue graft; test: collagen matrix) and 6 centers
Who Masked: Investigator, Outcomes Assessor
Masking Description: It concerns a surgical intervention. Hence, the treating surgeon and patient cannot be masked. The investigators and outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Connective tissue graft harvested from the palate
  Interventions: Procedure: Soft tissue augmentation at the buccal aspect of single implants
- Collagen matrix (Experimental): Pig-derived collagen matrix (Fibro-Gide, Geistlich Biomaterials, Wolhusen, Switserland)
  Interventions: Procedure: Soft tissue augmentation at the buccal aspect of single implants

INTERVENTIONS:
Procedure: Soft tissue augmentation at the buccal aspect of single implants — Soft tissue augmentation is performed following mucoperiosteal flap elevation at the buccal aspect of single implants. The connective tissue graft (control) or collagen matrix (test) is inserted in the buccal pouch and attached with monofilament sutures.

SUMMARY:
Patients in need of a single implant in the premaxilla and presenting with a horizontal buccal soft tissue defect at the single tooth gap will be invited to participate in a multicenter RCT. Prior to surgery, a small-field low-dose CBCT is taken since a buccopalatal bone dimension of at least 6 mm at the central and crestal aspect of the single tooth gap is required to ensure complete embedding of an implant by bone. Sixty patients will be randomly allocated to the test group or control group in 6 centers. Each center receives 10 sealed envelopes (5 are internally labelled with 'test group' and 5 with 'control group').

For each patient a digital planning is performed in implant planning software and a tooth-supported surgical guide is fabricated. In the control group, a single implant is placed following flap elevation and surgical guide installation. Then, a CTG from the palate is positioned under the buccal mucosa to thicken the tissues. A provisional restoration is placed at the day of surgery, which is replaced by a permanent one 3m later. Patients in the test group are treated in the same way, yet a CM (Fibro-Gide®) is used instead of a CTG.

Changes in the buccal soft tissue profile are registered over time by superimposing intra-oral scans in SMOP® software.

Secondary outcomes included clinical, aesthetic and patient-reported outcomes.

DETAILED DESCRIPTION:
Patients will be included in a multicenter RCT following screening and after having received written consent.

A sample size calculation using the Satterthwaite t-test was performed in SAS Power and Sample Size based on a comparison of mean change in BSP (primary outcome variable) from baseline to 1 year between the control group and test group. The calculation was based on finding a mean difference of at least 0.5 mm between these groups with a standard deviation of 0.5 mm for CTG and 0.7 mm for CM (as adopted from Zeltner et al. 2017). With alpha set at 0.05 and a power of 0.80, the sample size calculation indicated 25 patients to be included per group. To compensate for drop-outs, 30 patients would be treated with CTG and 30 would be treated with CM.

Clinicians and centers, randomization, allocation concealment and blinding Six experienced clinicians will treat 10 patients each. All clinicians are staff members of the Department of Periodontology and Oral Implantology at UGent - UZ Gent, who also work part-time in different private practices. The digital workflow, the implant placement protocol, the application of CTG and CM and the restorative protocol will be thoroughly discussed among the 6 clinicians in a training session before the start of the trial.

During the training session each clinician will receive 5 sealed envelopes internally coded as 'CTG' and another 5 as 'CM'. Just prior to surgery, a sealed envelope will be randomly selected and opened to reveal the treatment to be conducted. The measuring investigator will not be involved in the treatment of any of the patients and will be blinded to allow unbiased registrations.

Pre-operative digital planning A full digital workflow will be adopted for every patient. This implies the fabrication of a stereolythographic surgical guide on the basis of a 3D digital implant planning in designated software (NobelClinician, Nobel Biocare, Zürich, Switserland). A low-dose small-field Cone-Beam CT and intra-oral scan are required for this purpose. The same software will also be used to design a provisional acrylic crown, which will be adapted chairside immediately following surgery (Tempshell, Nobel Biocare, Zürich, Switserland).

Surgery Control group: soft tissue augmentation with CTG Patients start to take systemic antibiotics (Amoxicilline 1g) and anti-inflammatory medication (ibuprofen 600 mg) 1h pre-operatively. Following local anesthesia (Septanest special, Septodont, Saint Maur des Fossés, France) and oral disinfection (Corsodyl mouth rinse, GSK, Wavre, Belgium), a conventional mucoperiosteal flap will be raised. Thereupon, the surgical guide is positioned and a dental implant (NobelReplace CC PMC, Nobel Biocare, Zürich, Switserland) is installed. A CTG is harvested from the palatal mucosa in the premolar area by means of the single-incision technique as described by De Bruyckere et al. (2015) (fig. 1). The CTG is pulled into the envelope and fixed with two sutures (Seralon 6/0, Serag Weissner, Naila, Germany). Tension-free primary wound closure with the same suture material is pursued around a provisional acrylic crown. Post-op instructions include the intake of systemic antibiotics during 4 days (Amoxicilline 1g, two times a day), anti-inflammatory medication as deemed necessary by the patient and oral disinfection twice a day during 1 week. Then, sutures are removed. After 3 months, the provisional crown will be replaced by a permanent crown by the general dentist.

Test group: soft tissue augmentation with CM In the test group, no CTG is harvested as it will be replaced by CM (Fibro-Gide, Geistlich Biomaterials, Wolhusen, Switserland). Apart from that, all pre-op, surgical and post-op procedures are identical in the control group and test group.

Prior to surgery (baseline = t0), at 3 months (t1), 1 year (t2) and 5 years (t3) an intra-oral optical scan of the implant site and neighboring teeth will be taken (Trios, 3shape, Copenhagen, Denmark). The region of interest (ROI) will be defined on STL files with a trapezoid shape encompassing the following borders: 1 mm apical to the midbuccal soft tissue level (coronal), the mucogingival junction (apical) and 1 mm distance from the neighbouring tooth at both sides (mesial, distal). This ROI may vary between patients due to anatomical variation but will be kept constant in each patient and site over time. The STL images of baseline and follow-up will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. The linear changes in BSP will be measured in the middle of the ROI, calculated by the software and expressed in mm corresponding to the mean distance between the surfaces representing the evaluated time points (t0, t1, t2, t3).

All patients are scheduled for suture removal and oral hygiene instructions after 1 week with registration of:

Postoperative bleeding, Pain and amount of anti-inflammatory medication taken, Oedema and Hematoma.

After 3 months, 1 year and 2 years, all patients are scheduled for a clinical and radiographic follow-up visit, including registration of mesial and distal marginal bone level. Intra-oral radiographs will be taken using the long-cone parallel technique. Bone levels will be assessed and defined as the distance from the implant-abutment interface to the first bone-to-implant contact to the nearest 0.1 mm. Clinical parameters ,such as probing pockets depths (mm), plaque (presence or absence) and bleeding on probing (presence or absence) are registered as well as vertical soft tissue levels at the midbuccal aspect to the nearest 0.5 mm. White and Pink esthetics are assessed according to Furhauser.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* good oral hygiene defined as full-mouth plaque score ≤ 25%
* presence of a single tooth gap in the anterior maxilla (15-25) with both neighboring teeth present
* failing tooth at least 3 months earlier removed
* class I defect at the single tooth gap as clinically assessed (buccopalatal loss of tissue with a normal apicocoronal ridge height)
* buccopalatal bone dimension of at least 6 mm at the central and crestal aspect of the single tooth gap to ensure complete embedding of an implant by bone.

Exclusion Criteria:

* systemic diseases
* smoking
* (history of) periodontal disease;
* untreated caries lesions
* need for horizontal bone augmentation at the time of implant placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in buccal soft tissue profile (BSP) | Pre-op, 3 months, 1 year, 2 years
  Volumetric analysis with designated software on the basis of intra-oral scans at fixed time points (absolute changes in mm, relative changes in %)

SECONDARY OUTCOMES:
Changes in Probing pocket depth | 3 months, 1 year, 2 years
  Probing pocket depth (mm)
Changes in Bleeding on probing | 3 months, 1 year, 2 years
  Bleeding on probing (score 0-4)
Changes in Plaque Index | 3 months, 1 year, 2 years
  Plaque index (score 0-4)
Changes in radiographic outcomes | 3 months, 1 year, 2 years
  marginal peri-implant bone loss (mm)
Patient-reported outcome measures | 1 week
  Assessment of pain (VAS)
Patient-reported outcome measures | 1week
  oedema (VAS)
Patient-reported outcome measures | 1 week
  bleeding (VAS)
Patient-reported outcome measures | 1 week
  hematoma (VAS)
Patient-reported outcome measures | 1 week
  aesthetic evaluation by patients (VAS)
Patient-reported outcome measures | 3 months
  aesthetic evaluation by patients (VAS)
Patient-reported outcome measures | 1 year
  aesthetic evaluation by patients (VAS)
Patient-reported outcome measures | 2 years
  aesthetic evaluation by patients (VAS)
Patient-reported outcome measures | 1 week
  willingness to undergo again (VAS)
Patient-reported outcome measures | 3 months
  willingness to undergo again (VAS)
Patient-reported outcome measures | 1 year
  willingness to undergo again (VAS)
Patient-reported outcome measures | 2 years
  willingness to undergo again (VAS)
Aesthetic outcome as assessed by care providers | 1 year
  Pink Esthetic Score (0-14)
Aesthetic outcome as assessed by care providers | 2 year
  Pink Esthetic Score (0-14)
Aesthetic outcome as assessed by care providers | 1 year
  WhiteEsthetic Score (0-10)
Aesthetic outcome as assessed by care providers | 2 years
  White Esthetic Score (0-10)
Surgery time | At Surgery
  Time needed to complete the contour augmentation procedure
Primary stability | At Surgery
  Primary stability after implant placement (Ncm)
Incremental cost-effectiveness ratio | baseline - 2 years
  Difference in cost divided by the effect of the different procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be included in a meta-analysis upon request by the authors, they can be transferred

REFERENCES:
- [Background] Burkhardt R, Hammerle CH, Lang NP; Research Group on Oral Soft Tissue Biology & Wound Healing. Self-reported pain perception of patients after mucosal graft harvesting in the palatal area. J Clin Periodontol. 2015 Mar;42(3):281-7. doi: 10.1111/jcpe.12357. Epub 2015 Feb 16. PMID 25544993
- [Background] De Bruyckere T, Eeckhout C, Eghbali A, Younes F, Vandekerckhove P, Cleymaet R, Cosyn J. A randomized controlled study comparing guided bone regeneration with connective tissue graft to re-establish convexity at the buccal aspect of single implants: A one-year CBCT analysis. J Clin Periodontol. 2018 Nov;45(11):1375-1387. doi: 10.1111/jcpe.13006. PMID 30133718
- [Background] De Bruyckere T, Eghbali A, Younes F, De Bruyn H, Cosyn J. Horizontal stability of connective tissue grafts at the buccal aspect of single implants: a 1-year prospective case series. J Clin Periodontol. 2015 Sep;42(9):876-882. doi: 10.1111/jcpe.12448. Epub 2015 Sep 16. PMID 26373422
- [Background] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Background] Eghbali A, Seyssens L, De Bruyckere T, Younes F, Cleymaet R, Cosyn J. A 5-year prospective study on the clinical and aesthetic outcomes of alveolar ridge preservation and connective tissue graft at the buccal aspect of single implants. J Clin Periodontol. 2018 Dec;45(12):1475-1484. doi: 10.1111/jcpe.13018. Epub 2018 Nov 5. PMID 30290007
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307
- [Background] Huber S, Zeltner M, Hammerle CHF, Jung RE, Thoma DS. Non-interventional 1-year follow-up study of peri-implant soft tissues following previous soft tissue augmentation and crown insertion in single-tooth gaps. J Clin Periodontol. 2018 Apr;45(4):504-512. doi: 10.1111/jcpe.12865. Epub 2018 Feb 1. PMID 29290089
- [Background] Naenni N, Bienz SP, Benic GI, Jung RE, Hammerle CHF, Thoma DS. Volumetric and linear changes at dental implants following grafting with volume-stable three-dimensional collagen matrices or autogenous connective tissue grafts: 6-month data. Clin Oral Investig. 2018 Apr;22(3):1185-1195. doi: 10.1007/s00784-017-2210-3. Epub 2017 Sep 18. PMID 28924826
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Seibert JS. Reconstruction of deformed, partially edentulous ridges, using full thickness onlay grafts. Part I. Technique and wound healing. Compend Contin Educ Dent (Lawrenceville). 1983 Sep-Oct;4(5):437-53. No abstract available. PMID 6578906
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Thoma DS, Buranawat B, Hammerle CH, Held U, Jung RE. Efficacy of soft tissue augmentation around dental implants and in partially edentulous areas: a systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S77-91. doi: 10.1111/jcpe.12220. PMID 24641003
- [Background] Thoma DS, Naenni N, Benic GI, Hammerle CH, Jung RE. Soft tissue volume augmentation at dental implant sites using a volume stable three-dimensional collagen matrix - histological outcomes of a preclinical study. J Clin Periodontol. 2017 Feb;44(2):185-194. doi: 10.1111/jcpe.12635. Epub 2017 Jan 3. PMID 27716970
- [Background] Thoma DS, Zeltner M, Hilbe M, Hammerle CH, Husler J, Jung RE. Randomized controlled clinical study evaluating effectiveness and safety of a volume-stable collagen matrix compared to autogenous connective tissue grafts for soft tissue augmentation at implant sites. J Clin Periodontol. 2016 Oct;43(10):874-85. doi: 10.1111/jcpe.12588. Epub 2016 Aug 12. PMID 27310522
- [Background] Tonetti MS, Jepsen S; Working Group 2 of the European Workshop on Periodontology. Clinical efficacy of periodontal plastic surgery procedures: consensus report of Group 2 of the 10th European Workshop on Periodontology. J Clin Periodontol. 2014 Apr;41 Suppl 15:S36-43. doi: 10.1111/jcpe.12219. PMID 24640999
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Zeltner M, Jung RE, Hammerle CH, Husler J, Thoma DS. Randomized controlled clinical study comparing a volume-stable collagen matrix to autogenous connective tissue grafts for soft tissue augmentation at implant sites: linear volumetric soft tissue changes up to 3 months. J Clin Periodontol. 2017 Apr;44(4):446-453. doi: 10.1111/jcpe.12697. Epub 2017 Feb 11. PMID 28107560
- [Background] Zucchelli G, Mounssif I, Mazzotti C, Montebugnoli L, Sangiorgi M, Mele M, Stefanini M. Does the dimension of the graft influence patient morbidity and root coverage outcomes? A randomized controlled clinical trial. J Clin Periodontol. 2014 Jul;41(7):708-16. doi: 10.1111/jcpe.12256. Epub 2014 May 8. PMID 24708394
- [Derived] Surdiacourt L, Christiaens V, De Bruyckere T, De Buyser S, Eghbali A, Vervaeke S, Younes F, Cosyn J. A multi-centre randomized controlled trial comparing connective tissue graft with collagen matrix to increase soft tissue thickness at the buccal aspect of single implants: 3-Year results. J Clin Periodontol. 2025 Jan;52(1):92-101. doi: 10.1111/jcpe.13975. Epub 2024 Mar 14. PMID 38485651
- [Derived] Cosyn J, Eeckhout C, De Bruyckere T, Eghbali A, Vervaeke S, Younes F, Christiaens V. A multi-centre randomized controlled trial comparing connective tissue graft with collagen matrix to increase soft tissue thickness at the buccal aspect of single implants: 1-year results. J Clin Periodontol. 2022 Sep;49(9):911-921. doi: 10.1111/jcpe.13691. Epub 2022 Jul 20. PMID 35781692
- [Derived] Cosyn J, Eeckhout C, Christiaens V, Eghbali A, Vervaeke S, Younes F, De Bruyckere T. A multi-centre randomized controlled trial comparing connective tissue graft with collagen matrix to increase soft tissue thickness at the buccal aspect of single implants: 3-month results. J Clin Periodontol. 2021 Dec;48(12):1502-1515. doi: 10.1111/jcpe.13560. Epub 2021 Oct 12. PMID 34605057